CLINICAL TRIAL: NCT02135588
Title: Combination Tissue Plasminogen Activator (Tpa) and Dornase Alfa (Dnase) Administration Through Intrapleural Catheters for the Treatment of Loculated or Non-Draining Malignant Pleural Effusions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERMC 13-29
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Loculated or Non-draining Malignant Pleural Effusions
MeSH Terms: interventions — dornase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Treatment (Experimental): Intra-pleural deoxyribonuclease 5mg and intra-pleural Alteplase 10mg, every 12 hours over 72 hours (total of 6 treatments)
  Interventions: Drug: Combination TISSUE PLASMINOGEN ACTIVATOR (TPA) AND DORNASE ALFA (DNASE)

INTERVENTIONS:
Drug: Combination TISSUE PLASMINOGEN ACTIVATOR (TPA) AND DORNASE ALFA (DNASE)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intrapleural dornase alfa and tPA administered to patients with clinical failure of small-bore chest tube with persistent pleural effusions or malignancy-related loculated effusion to improve pleural drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical failure of small-bore chest tube with persistent pleural effusion
2. 18 years of age or older
3. Eastern Cooperative Oncology Group (ECOG) performance status score 0-2.
4. Life expectancy ≥ 6 weeks
5. Absolute neutrophil count > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 8.0 g/dL
6. Serum creatinine ≤2.0 times the upper limit of the normal range, total bilirubin ≤ 2.5 mg/dL, AST/ALT ≤ 5 times the upper limit of normal range
7. At least 2 days from administration of chemotherapy
8. At least 7 days from prior major surgery
9. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial.
10. Patient judged to be 'medically stable' by primary investigator.

Exclusion Criteria:

1. Prior treatment with intrapleural fibrinolytic agents
2. Presence of any intracranial mass
3. Traumatic hemorrhagic pleural effusion
4. Major hemorrhage, coincidental stroke, or major trauma
5. High-risk for systemic bleeding
6. Allergy or intolerance to dornase alfa
7. Active clinically serious infection > CTCAE (version 4.03) Grade 2.
8. Serious non-healing wound, ulcer, or bone fracture.
9. Major surgery, open biopsy or significant traumatic injury within seven (7) days of first study drug--including neurosurgery.
10. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements.
11. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements.
12. Patients who are pregnant or lactating (females of childbearing potential must have a negative pregnancy test prior to participation in this study)
13. Expected survival less than six weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic improvement in area of pleural collection | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Steven B Standiford, MD, Principal Investigator — Eastern Regional Medical Center, Inc.
Locations (1):
- Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States